CLINICAL TRIAL: NCT03231462
Title: Impact of Perioperative Physical Activity on Postoperative Pulmonary Complications and Quality of Life Among Esophageal Cancer Patients: A Prospective Cohort Study
Brief Title: Impact of Perioperative Physical Activity on Postoperative Pulmonary Complications and Quality of Life Among Esophageal Cancer Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Samsung Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: 2014-10-035
Record Dates: First submitted 2017-07-10; First posted 2017-07-27 (Actual); Last update posted 2018-10-11 (Actual); Status verified 2018-09

CONDITIONS: Esophageal Neoplasms
MeSH Terms: conditions — Esophageal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This prospective cohort study examines the impact of perioperative physical activity on postoperative pulmonary complications among esophageal cancer patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are diagnosed with esophageal cancer and scheduled to receive curative esophagectomy
* Patients who are able to read and understand the questionnaire
* Patients who are able to communicate with research personnel
* Patients who recognize the purpose of this study and provide written informed consent
* Patients without treatment for psychiatric disease

Exclusion Criteria:

* Patients who have difficulty for walking
* Patients with history of other cancer in the last 3 years
* Patients with neoadjuvant chemotherapy and/or radiation therapy
* Patients with recurrent esophageal cancer
* Patients with multiple cancer
* Foreigner or overseas patients who were not able to regularly participate this study

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who are diagnosed with eshophageal cancer and scheduled to receive curative esophagectomy at a single cancer hospital in Seoul, Korea
Sampling Method: Probability Sample
Enrollment: 180 (Estimated)
Dates: Start 2015-03-06 (Actual); Primary Completion 2019-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Pulmonary complications | Within 30 days after surgery
  Incidence of pneumonia and atelectasis

SECONDARY OUTCOMES:
The change of quality of life | Before surgery(baseline), and 1, 6, 12, 24, 36, 48, and 60 months after surgery
  The change of quality of life is measured using the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire (EORTC QLQ) core30 (C30). The quality of life scale is transformed into a score 0 to 100, derived by 4-point Likert scale. A higher score represents a higher level of quality of life.
The change of symptom | Before surgery(baseline), and 1, 6, 12, 24, 36, 48, and 60 months after surgery
  The change of symptoms is measured using the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire (EORTC QLQ) oesophageal cancer module (OES18). The symptom scale is transformed into a score 0 to 100, derived by 4-point Likert scale. A higher score represents a higher level of symptom.

CONTACTS AND LOCATIONS:
Overall Officials: Young Mog Shim, MD, Principal Investigator — Samsung Medical Center
Locations (1):
- Samsung Medical Center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No